CLINICAL TRIAL: NCT04188470
Title: Open Randomised Multicentric Controlled Trial to Evaluate the Impact of an Intervention to Improve Drug Appropriateness in Polymedicated Patients According to the Person-centered Care Model by a Multidisciplinary Team At Primary Care
Brief Title: Optimising Drug Therapy in Polymedicated Patients According to the Person-centered Care Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19/144-P
Record Dates: First submitted 2019-12-03; First posted 2019-12-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Multiple Chronic Conditions; End Stage Disease
Keywords: Polypharmacy; deprescriptions; patient-centered care; frail elderly; interprofessional relations; decision making
MeSH Terms: conditions — Multiple Chronic Conditions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- person-centered care model (Experimental): healthcare multidisciplinary team will review the appropriateness of medication by a person-centered care model and then the healtcare team will propose changes in the therapeutic plan to the patient or caregiver
  Interventions: Behavioral: person-centered care model
- usual care (No Intervention): the healthcare team will practice usual care

INTERVENTIONS:
Behavioral: person-centered care model — A multidisciplinary team (clinical pharmaceutical, expert physician on chronic management disease, and basic healthcare team) will review the frailty, complexity, the therapeutic goals of the patients to propose changes on the therapeutic plan to improve the appropriateness, these changes will we agreed with the patient or caregiver.
  Arms: person-centered care model

SUMMARY:
Introduction: In recent years, multi-aging has increased by 25%. This is related to plutipatology, frailty, polymedications, elevated sanitary cost, low quality of life, adverse events and mortality. To improve this it is necessary to apply the people-centered care model that includes and individualized therapeutic plan taking into account medication appropriateness, frailty, complexity and patient preferences. A collaborative model by a multidisciplinary team is proposed to make decisions to optimize drug therapy.

Hypothesis: person-centered care model by a multidisciplinary team at primary care improve drug appropriateness in polymedicated elderly patients Material and Method: Design: Randomized (1:1), open-label, multicentre, parallel-arm clinical trial with 1-year follow-up. Study population: community-dwelling polymedicated (≥8 drugs) elderly (≥75 years old) people at 11 primary healthcare team in Bages, Osona and Anoia (Catalonian region). Period: May 2020 and ends at 12 months of follow-up of the last included subject. Method: 11 primary healthcare team will be randomized to control or intervention group, then volunteers basic healthcare team will participate in the study and they will be assigned to control or intervention group depending on which team they work, then the subjects assigned to theses basic healthcare teams that meet the inclusion criteria and not exclusion criteria will be selected and finally the informed consent of these will be obtained. In the intervention group the multidisciplinary work team comprised by the clinical pharmacist, expert collaborator doctor and the basic healthcare team will meet periodically to review subjects, a multidimensional review will be carried out by assessing the frailty, complexity, morbidity and the appropriateness drug therapy, if proposed changes in the therapeutic plan will have to be agreed with the patient taking into account their preferences. At 6 and 12 months or when their basic healthcare team requests it they will be reviewed again. In the control group the necessary study data collection will be carry out at the beginning and at 6 and 12 months, and the routine clinical practice in relation to the use of medication will be carried out. Measurements: variation of the mean of incidents (potencially prescription inadequate) per patient, variation of the number of prescribed drugs per patient, changes in the therapeutic plans implemented and variation of the number of hospitalizations.

DETAILED DESCRIPTION:
JUSTIFICATION:

The proposed project focuses on the clinical review from primary care because the healthcare team are close to the community-dwelling people and therefore offer integral care. The added value is given by the participation of a multidisciplinary team, in addition to the reference healthcare team, an expert chronicity physician and the primary care pharmacist are also involved, thus offer a greater amplitude in the centered vision and care in the patient and in the process of therapeutic appropriateness.

The Primary Care Pharmacist (FAP) in the Project ENAPISC, defined in Catalonia, positions itself as a necessary healthcare professional in the healthcare teams to ensure adequacy use of the medication.

Although the evidence published on the result of the implementation of these interventions in the primary care environment is multiple, its application is still scarce, which gives added value to the realization of the project.

OBJECTIVES:

GENERAL: To evaluate the effectiveness of the intervention to improve the therapeutic appropriateness of the elderly polymedicated patients by the application of person-centered prescription review method.

SPECIFIC:

* Describe the characteristics of the sample
* Decrease the number of detected incidents in the prescription
* Decrease the number of prescribed medications
* -decrease the numer of hospitalizations
* Detect if there are incidents related to the medication derived from the intervention done.
* Know the changes produced in the medication plan of the intervention group after one year after the intervention has finished.

METHODS:

Study design: Randomized (1:1), open-label, multicentre, parallel-arm clinical trial with 1-year follow-up Study period: May 2020-May 2024. Study population: polymedicated patients with the condition of complex chronic patient or patient with advanced chronic disease and / or ≥ 75 years old assigned to 11 primary healthcare teams in Bages, Osona and Anoia.

Selection of the primary care center, the basic healthcare team and the subjects: Of the 11 primary care center that belong to the scope of work of the FAP, volunteer basic healthcare team will participate, these will be randomized and then the possible subjects that meet the criteria of the study population are selected, taking into account the inclusion and exclusion criteria with the calculation of the size of the study population and the sampling procedure we obtain the selection of participants.

Randomization and distribution of subjects: the 11 primary care team will be graded in a 1:1 proportion, then basic healthcare team will be assigned to control or intervention group depending on which team they will work, to prioritize study subjects, those that are in the list of possible subjects will be selected, and finally the informed consent will be obtained. It is an open study, therefore, the subjects and the basic healthcare team will be aware of what group of study they belong to.

Sample size and sampling procedure:

The sample size has been calculated using the GRANMO v.7.12 program for two independent proportions. With an alpha risk of 0.05, a beta of 0.20 with a loss ratio of 0.15.

146 subjects are needed in the first group and 146 in the second group to detect how statistically significant the difference between two proportions of the average reduction in the number of medications per patient, which for group 1 is expected to be 0.23 and for group 2 of 0.10 . Approximation of ARCSINUS has been used.

Collection of data and sources of information:

The list of patients defined as study population and who meet criteria of inclusion and no exclusion criteria will be requested from the information systems of the company, the subjects will be recruited through a telephone visit and in case of acceptance of the participation the subjects must sign the informed consent that will be offered to them through a visit with nursing to the center or at home if necessary. The control group or the intervention group will be assigned according to the basic healthcare team to which they are assigned.

The data necessary to carry out the study and defined in the data collection sheets, should be obtained from electronic clinical history.

Data analysis:

A description of the variables will be made by calculating proportions in the case of qualitative variables and representation with the corresponding graphs and a median calculation in the case of normal or median distribution if this is not the case for quantitative variables.

Bivariate inferential analysis with a parametric test in the case of normal distribution of comparison of means (t-STUDENT), and in the case of non-normal distribution a non-parametric equivalent test, in particular, the Mann-Whitney U will be used. And in the case of comparison between categorical variables we will use the Ji-cuadrado to determine the relation between variables and the Cramer V test to determine the intensity of the association in case there is one.

Multiple regression to analyze the effect of the confusing variables on the main result variable.

The statistical program SPSS v24.0 will be used to analyze the data.

WORK PLAN:

Basic healthcare team will be randomized and the subjects of study will be control or intervention depending on the assigned basic healthcare team.

In the intervention group, the work group formed by the primary care pharmacist and the physician and nurse assigned to the patients, will meet periodically to analyze 2-4 patients each meeting, a multidimensional patient review will be carried out to evaluate the frailty, complexity, health problems, control of clinical variables to assess the appropriateness of the medication by means of the detection of incidents, the group will propose changes in the therapeutic plan which will have to be finally agreed with the patient or caregiver. They will be reviewed again at 6 and 12 months. Nursing will schedule visit 0 with the patient or caregiver and the data be collected. At the same time, in a bi-annual manner, meetings with the work group will be scheduled. Once reviewed the basic healthcare team will schedule visits with the patient:

* Visit 1 to 15 days after the group meeting
* visit at 3 months to keep track of agreed changes
* Visit at 6 and 12 months prior to the work group meeting about 15 days before In the case of need for support from the community pharmacist or the social worker or other physicians, an individualized work plan will be agreed with them.

At 6 months or earlier, if a member of the group requires it, the patient's therapeutic plan will be reviewed again to monitor the clinical follow-up of the patient, to review whether there has been any incidence in the therapeutic plan adaptation process, and / or make more changes.

In the subjects of the control group the necessary data will be collected to carry out the study at the beginning and at 6 and 12 months, and the usual clinical practice will be done in relation to the use of medication. Nursing will program 3 visits (0, 6 and 12 months) in the center or at home to perform data collection, and the pharmaceutical will review the therapeutic plan.

Finally, the data of each patient included in the study will be introduced on the file created to track and evaluate results.

DIFFICULTIES AND LIMITATIONS OF THE STUDY:

The beliefs of healthcare professionals who treat patients may make it difficult to improve the adaptation of the therapeutic plan but it is considered that the design of the project (randomized trial), the multidisciplinary team work, the participation of an expert in the use of the medication can help reduce the impact of this factor and redirect some beliefs; The management of the time is also a limitation because the exhaustive review of the patient's therapeutic plan requires some time, but in this case, the health benefit that the project can generate can make the investment of time efficient. The results can be biased by the effect of the professionals on the control group and on the part of the patients knowing that they participate in the study (open study). Finally, the knowledge and beliefs of patients regarding medication and health can also be a factor that hinders changes in the therapeutic plan but with an appropriate process of shared decisions where quality information is worked for the patient, the autonomy and the decision-making capacity may reduce the impact of this limitation.

APPLICABILITY AND PRACTICAL USE OF THE RESULTS:

The proposed model proposes a systematic work in the process of medication review and teamwork with the approach from different points of view and degrees of knowledge of the subject. Until now, the medication review is done without applying a systematic process and without taking into account the technical knowledge of other skilled professionals.

Considering as a general and last objective to improve the therapeutic appropriateness of polymedicated patients, this is an innovative model, since it is characterized by:

* multidisciplinary team work: each professional provides different knowledge and perspectives regarding the use of the medication and the patient's knowledge, and the sum of all contributes the added value of the person-centered care model.
* incorporation of the primary care pharmacist as a reference in the safe and quality use of the medication in the person-centered care assistance process.

ETHICAL ASPECTS:

The project will be presented to the Committee of Ethics and Research (CEI) of the IDIAP and the Bioethics Committee of the University of Barcelona (CBUB) to request approval.

The project will be explained to the patients selected, the patient information sheet will be delivered, and the informed consent will be requested to participate in the study, which must be signed. In the case of a patient with moderate-advanced dementia the consent of both patients and caregivers will be required, and in the case of an invalid patient the consent must be signed by the legal guardian.

The participation in the investigation is voluntary and the subjects will be able to exercise the rights of access, rectification, suppression, right to the limitation of the treatment, as well as to the portability and opposition, whenever the exercise of these rights does not affect the purposes of the investigation.

The ethical principles for biomedical research on human subjects are fulfilled. In accordance with the provisions of Organic Law 3/2018, of December 5, on the protection of personal data and the guarantee of digital rights, personal information will always be treated through codes. The information recorded is encrypted for transfer to the database of the study. All servers have antivirus protection, firewalls, controlled access, permanent surveillance, alarms, as well as other relevant security measures to ensure the protection of information.

The study will generate several files with personal data. These will be kept only for the duration of the study and will be stored under the custody of the principal investigator in the directory of the shared unit of the company where she's working (SAPDIRASSIST \ Medication Area \ CAROL ROVIRA \). However, these files will be password protected despite being stored in a private directory. The data collected already consists of the authorization of the people whose data will be part of this study, complying with the applicable laws on data protection (LOPD-GDD and RGPD).

The subjects of the study may exercise their rights of access, rectification, deletion, right to limit the treatment of their data, as well as portability and opposition, provided that the exercise of these rights does not affect the purposes of investigation for which they were collected.

ELIGIBILITY:
Inclusion Criteria:

* Polimedicated patients (>7 drugs of >1 month treatment duration, exclude topical drugs, ophtalmologic drugs, diaper and cure products)
* Multiple chronic conditions
* Advanced cronic disease with short life expectancy

Exclusion Criteria:

* Subjects do not want participate at the study
* <2 visits in the last year with the basic healthcare team
* palliative care by PADES

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 208 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
average number ofdetected incidents | 0 and 12 months
  Medication incidents defined as therapeutic duplicity, contraindications, security advice about a drug, avoidable medication, inadequate duration, combinations of anticholinergic drugs, medication not recommended in older people, inadequate dosage, drug more efficient, and medication not indicated.
average on number of drugs per patient | 0 and 12 months
  number of chronic (>1 month of treatment duration) drugs (excluded topic drugs, ophthalmic drugs, diapers and cure material) prescribed in the therapeutic plan of the patient
average of medication changes | 6 and 12 months
  number of changes maked in the therapeutic plan of the patients
average of hospitalizations | 0 and 12 months
  number of hospitalizations

SECONDARY OUTCOMES:
Number of adverse events caudes by medication changes | 6 and 12 months
  Adverse events caused by the intervention defined as abstinence syndrome, rebound effects, worsening symptoms, medication errors, emergency visitors, hospital admissions, successes
Number of changes at the end of the study | 6 and 12 months
  Medication changes at th end of the study define as a reintroduction of a stopped medication during the intervention and/or introduction of a new medication

CONTACTS AND LOCATIONS:
Overall Officials: Carol Rovira, Principal Investigator — ICS; Joan Armengol, Study Chair — ICS
Locations (2):
- Spain (2):
  - Mar Casanovas, Igualada, Barcelona
  - Rovira, Manresa, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodriguez-Manas L, Rodriguez-Artalejo F, Sinclair AJ. The Third Transition: The Clinical Evolution Oriented to the Contemporary Older Patient. J Am Med Dir Assoc. 2017 Jan;18(1):8-9. doi: 10.1016/j.jamda.2016.10.005. Epub 2016 Nov 22. No abstract available. PMID 27887892
- [Background] Campins L, Serra-Prat M, Gozalo I, Lopez D, Palomera E, Agusti C, Cabre M; REMEI Group. Randomized controlled trial of an intervention to improve drug appropriateness in community-dwelling polymedicated elderly people. Fam Pract. 2017 Feb;34(1):36-42. doi: 10.1093/fampra/cmw073. Epub 2016 Sep 7. PMID 27605543
- [Background] Melzer D, Tavakoly B, Winder RE, Masoli JA, Henley WE, Ble A, Richards SH. Much more medicine for the oldest old: trends in UK electronic clinical records. Age Ageing. 2015 Jan;44(1):46-53. doi: 10.1093/ageing/afu113. Epub 2014 Aug 7. PMID 25103030
- [Background] Yarnall AJ, Sayer AA, Clegg A, Rockwood K, Parker S, Hindle JV. New horizons in multimorbidity in older adults. Age Ageing. 2017 Nov 1;46(6):882-888. doi: 10.1093/ageing/afx150. PMID 28985248
- [Background] Bonaga B, Sanchez-Jurado PM, Martinez-Reig M, Ariza G, Rodriguez-Manas L, Gnjidic D, Salvador T, Abizanda P. Frailty, Polypharmacy, and Health Outcomes in Older Adults: The Frailty and Dependence in Albacete Study. J Am Med Dir Assoc. 2018 Jan;19(1):46-52. doi: 10.1016/j.jamda.2017.07.008. Epub 2017 Sep 9. PMID 28899661
- [Background] Onder G, Petrovic M, Tangiisuran B, Meinardi MC, Markito-Notenboom WP, Somers A, Rajkumar C, Bernabei R, van der Cammen TJ. Development and validation of a score to assess risk of adverse drug reactions among in-hospital patients 65 years or older: the GerontoNet ADR risk score. Arch Intern Med. 2010 Jul 12;170(13):1142-8. doi: 10.1001/archinternmed.2010.153. PMID 20625022
- [Background] Saum KU, Schottker B, Meid AD, Holleczek B, Haefeli WE, Hauer K, Brenner H. Is Polypharmacy Associated with Frailty in Older People? Results From the ESTHER Cohort Study. J Am Geriatr Soc. 2017 Feb;65(2):e27-e32. doi: 10.1111/jgs.14718. Epub 2016 Dec 26. PMID 28024089
- [Background] Hanlon JT, Schmader KE, Samsa GP, Weinberger M, Uttech KM, Lewis IK, Cohen HJ, Feussner JR. A method for assessing drug therapy appropriateness. J Clin Epidemiol. 1992 Oct;45(10):1045-51. doi: 10.1016/0895-4356(92)90144-c. PMID 1474400
- [Background] Spinewine A, Schmader KE, Barber N, Hughes C, Lapane KL, Swine C, Hanlon JT. Appropriate prescribing in elderly people: how well can it be measured and optimised? Lancet. 2007 Jul 14;370(9582):173-184. doi: 10.1016/S0140-6736(07)61091-5. PMID 17630041
- [Derived] Rovira C, Casanovas M, Vizcaino E, Massanes M, Miro Q, Sola L, Gallego J, Armengol J, Ayala C, Pascual J, Marino EL, Vidal-Alaball J, Modamio P; PCMR Study Group. Effectiveness of person-centred versus usual care in elderly patients: findings from a multicentre randomised controlled trial. J Pharm Policy Pract. 2026 Jan 19;19(1):2609020. doi: 10.1080/20523211.2025.2609020. eCollection 2026. PMID 41567179
- [Derived] Rovira C, Modamio P, Pascual J, Armengol J, Ayala C, Gallego J, Marino EL, Ramirez A; PCMR (Person-Centred Medication Review) Study Group. Person-centred care provided by a multidisciplinary primary care team to improve therapeutic adequacy in polymedicated elderly patients (PCMR): randomised controlled trial protocol. BMJ Open. 2022 Feb 9;12(2):e051238. doi: 10.1136/bmjopen-2021-051238. PMID 35140146
- See also: demographic data of catalonian population — https://www.idescat.cat/pub/?id=inddt&n=915&m=m
- See also: a guideline about drug selection at nursery homes — http://farmageriatrics.wordpress.com/guia-farmacoterapeutica/
- See also: document with definitions about chronic conditions — http://www.termcat.cat/ca/Diccionaris_En_Linia/160/Cerca/
- See also: document of catalonian health department about safe use of drugs — http://medicaments.gencat.cat/ca/professionals/seguretat/seguretat-clinica-recepta-electronica/
- See also: medication safe national institute — http://www.ismp-espana.org/estaticos/view/20
- See also: recommendations about clinical assessment and management in multimorbidity condition — http://www.nice.org.uk/guidance/ng56/chapter/Recommendations